CLINICAL TRIAL: NCT01640275
Title: The Effect of Isoflurane Versus Propofol Anesthesia on Alzheimers Disease CSF Markers
Brief Title: Markers of Alzheimers Disease After Propofol or Isoflurane Anesthesia
Acronym: MAD-PIA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00030861
Record Dates: First submitted 2012-06-20; First posted 2012-07-13 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-03

CONDITIONS: General Anesthesia
Keywords: General Anesthesia; Alzheimers Disease; Cognitive decline
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Propofol; Isoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol based intravenous anesthesia (Active Comparator): patients will receive propofol based intravenous anesthesia
  Interventions: Drug: Propofol
- Isoflurane Based Inhaled Anesthesia (Experimental): patients will receive isoflurane based inhaled anesthesia
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Propofol — patients randomized to the propofol arm of the study will receive general anesthesia with propofol
  Arms: Propofol based intravenous anesthesia
Drug: Isoflurane — patients randomized to the isoflurane arm of the study will receive general anesthesia with isoflurane
  Arms: Isoflurane Based Inhaled Anesthesia

SUMMARY:
Previous work in animal models suggests that inhalational anesthetic agents may accelerate Alzheimer's disease pathogenesis, but it is unclear to what extent this may happen in humans. Here, the investigators propose to measure Alzheimer's disease-related neural markers in the cerebrospinal fluid (CSF) of patients exposed to anesthesia while undergoing neurosurgical procedures that require lumbar drain placement. Patients will be randomized to either receive inhalation anesthesia with isoflurane or intravenous anesthesia with propofol.

CSF and blood samples will each be collected at the induction of anesthesia, and then again ten and twenty-four hours later. CSF samples will be assayed for amyloid beta, tau, and other Alzheimer's disease-associated markers; blood samples will be assayed for serum inflammatory markers and used for genotyping studies. These studies should clarify the effect of common anesthetic agents on Alzheimer's disease related neural markers.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and above
* seen in neurosurgical clinic, and scheduled for operative aneurysm repair or other neurosurgical procedure necessitating lumbar drain placement.
* ability to speak English.
* ability to understand consent forms, and to give informed consent.

Exclusion Criteria:

* age less than 18
* lumbar drain is not placed
* not eligible for one of the anesthetics (inhaled isoflurane or IV propofol)
* inmate of a correctional facility (i.e. prisoners).
* pregnancy. Pregnancy is ruled out as standard of care before cranial surgery, based on clinical history and/or HCG testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2012-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Ratio of cerebrospinal fluid tau to amyloid beta | twenty four hours after the induction of anesthesia

SECONDARY OUTCOMES:
the relationship between anesthetic exposure and CSF biomarker changes | up to 24 hrs after induction of anesthesia
the relationship between anesthetic exposure and CSF biomarker changes, and demographics (age, gender, and race) | up to 24 hrs after induction of anesthesia
the relationship between CSF biomarker changes and serum markers of metabolic and/or inflammatory status | up to 24 hrs after induction of anesthesia
the relationship between anesthetic exposure and biomarker changes and serum markers of metabolic and/or inflammatory status | up to 24 hrs after induction of anesthesia
the relationship between anesthetic exposure and biomarker changes and neuroimaging results obtained as dictated by routine standard of care | up to 24 hours after induction of anesthesia
the relationship between anesthetic exposure and biomarker changes and depth of anesthesia, based on average BIS (bispectral index) monitoring signal | up to 24 hours after induction of anesthesia
the relationship between anesthetic exposure and biomarker changes and the time of day that surgery is performed | up to 24 hours after induction of anesthesia
the relationship between anesthetic exposure and biomarker changes with genetic polymorphisms in ApoE (apolipoprotein E) and other genes related to inflammation, metabolism, brain function and/or Alzheimer's disease | up to 24 hours after induction of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Miles Berger, MD, PhD, Principal Investigator — Duke University Medical Center, Department of Anesthesiology; Michael L James, MD, Principal Investigator — Duke University Medical Center, Department of Anesthesiology; David McDonagh, MD, Principal Investigator — Duke University Medical Center, Department of Anesthesiology
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Berger M, Ponnusamy V, Greene N, Cooter M, Nadler JW, Friedman A, McDonagh DL, Laskowitz DT, Newman MF, Shaw LM, Warner DS, Mathew JP, James ML; MAD-PIA Investigators. The Effect of Propofol vs. Isoflurane Anesthesia on Postoperative Changes in Cerebrospinal Fluid Cytokine Levels: Results from a Randomized Trial. Front Immunol. 2017 Nov 13;8:1528. doi: 10.3389/fimmu.2017.01528. eCollection 2017. PMID 29181002
- [Derived] Berger M, Nadler JW, Friedman A, McDonagh DL, Bennett ER, Cooter M, Qi W, Laskowitz DT, Ponnusamy V, Newman MF, Shaw LM, Warner DS, Mathew JP, James ML; MAD-PIA trial team. The Effect of Propofol Versus Isoflurane Anesthesia on Human Cerebrospinal Fluid Markers of Alzheimer's Disease: Results of a Randomized Trial. J Alzheimers Dis. 2016 Apr 15;52(4):1299-310. doi: 10.3233/JAD-151190. PMID 27079717